CLINICAL TRIAL: NCT04273191
Title: An Evaluation of Multimodal Neuroimaging Parameters in Women With Postpartum Depression Who Are Receiving ZULRESSO
Brief Title: A Study to Evaluate Multimodal Neuroimaging Parameters in Women With Postpartum Depression Who Are Receiving ZULRESSO™ (Brexanolone)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sage Therapeutics has decided not to proceed with this study at this time
Sponsor: Sage Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 547-EXM-401
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Postpartum Depression
Keywords: Postpartum Depression; ZULRESSO
MeSH Terms: conditions — Depression, Postpartum | interventions — brexanolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brexanolone (Experimental): Participants will receive a single dose of commercial brexanolone as part of standard of care.
  Interventions: Drug: Brexanolone

INTERVENTIONS:
Drug: Brexanolone — Brexanolone will be initiated and administered per the USPI and the associated REMS.
  Other Names: ZULRESSO™; SAGE-547

SUMMARY:
In this Phase 4 study, women who have been prescribed commercial ZULRESSO™ (brexanolone) by a physician as standard of care for postpartum depression (PPD) and who are planning to receive the infusion per United States Prescribing Information (USPI) at a Risk Evaluation and Mitigation Strategy (REMS)-certified healthcare center are being asked to participate to collect data on multimodal neuroimaging parameters in order to evaluate the relationship between changes in depressive symptoms and changes in neuroimaging parameters.

ELIGIBILITY:
Inclusion criteria:

* Participant has been prescribed brexanolone for PPD and plans to receive commercially available brexanolone per the USPI at a REMS-certified healthcare setting.
* Participant is ambulatory.
* Participant agrees to adhere to the study requirements.
* Participant has had a major depressive episode that began no earlier than the third trimester and no later than the first 4 weeks following delivery, as diagnosed by the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders (SCID-5).
* Participant agrees not to be the primary caregiver of any dependents during the infusion.
* Participant has a HAM-D total score of ≥22 at screening and baseline.
* Participant is ≤12 months postpartum at screening.
* Participant is willing at screening to delay the start of any new pharmacotherapy regimens, including antidepressant or antianxiety medication until the brexanolone infusion and post-Infusion assessments have been completed. If medically justified, any new medication should be delayed until after the Day 30 follow-up visit.
* If the participant is taking medications administered to treat the symptoms of depression or anxiety (such as anxiolytics or antidepressants), these must be at a stable dose from 30 days prior to dosing until the brexanolone infusion and post-infusion assessments have been completed. If medically justified, any change of preexisting medication should be delayed until after the Day 30 follow-up visit.
* Participant agrees to use a highly effective method of contraception during participation in the study and for 30 days following the end of the brexanolone infusion, unless she is surgically sterile (bilateral salpingectomy, bilateral oophorectomy, and/or hysterectomy) or does not engage in sexual relations which carry a risk of pregnancy.

Exclusion criteria:

* Participant has a positive pregnancy test at screening or baseline.
* Participant's most recent pregnancy resulted in a miscarriage, still birth, or neonatal death; or participant has terminated parental rights (eg, child has been placed for adoption).
* Participant has evidence of any gross brain abnormality observed during the baseline MRI, as determined by a radiologist.
* Participant has clinically significant findings considered to interfere with the participant's ability to safely participate in the study, as determined by the investigator upon evaluation of medical history, electrocardiogram, hematology, and clinical chemistry.
* Participant has end stage renal disease.
* Participant is in hepatic failure.
* Participant has known allergy to progesterone or allopregnanolone.
* Participant has active psychosis per investigator assessment.
* Participant has attempted suicide during the current episode of PPD.
* Participant has a medical history of bipolar disorder, schizophrenia, and/or schizoaffective disorder.
* Participant has current/active alcohol or drug abuse (including benzodiazepines) within the 30 days prior to screening as assessed by the investigator. A positive urine drug screen is exclusionary unless deemed by the investigator to reflect a prescribed medication.
* Participant has been exposed to an investigational medication or device within 30 days prior to screening.
* During the current episode of PPD, participant has participated in this study or any other study employing brexanolone, SAGE-217, ganaxolone, or a similar compound, or has received prior treatment with ZULRESSO™.
* Participant is investigative site personnel, sponsor personnel, or an immediate member of their family (spouse, parent, child, or sibling, whether biological or legally adopted).
* Participant has received electroconvulsive therapy within 30 days prior to screening and/or plans to receive electroconvulsive therapy before the Day 30 visit.
* MRI is contraindicated for the participant for any reason, including but not limited to: cardiac pacemaker, surgical implants, previous accident resulting in metal or shrapnel lodged internally, tattoos inked with metallic dyes, a history of metal work without using protective eyewear, history of claustrophobia.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Post-Infusion on the 17-item Hamilton Rating Scale for Depression (HAM-D) Total Score | Up to approximately 5 days
  The HAM-D total score comprises a sum of 17 individual item scores. Items scored in a range of 0 to 2 include: insomnia (early night, middle night, early morning), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. Items scored in a range of 0 to 4 include: agitation, depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The total score can range from 0 to 52.
Change from Baseline to Post-Infusion in Functional Connectivity Using Blood Oxygenation Level-Dependent (BOLD) Resting State Functional Magnetic Resonance Imaging (rsfMRI) | Up to approximately 5 days
  rsfMRI is used in brain mapping to evaluate regional interactions that occur in a resting or task-negative state, when an explicit task is not being performed.

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.